CLINICAL TRIAL: NCT04566094
Title: Lung Herniation After Uniportal VATS. Rarity or Common Finding?
Brief Title: Lung Herniation After Uniportal VATS
Status: Withdrawn | Type: Observational
Why Stopped: PIs moved to other department
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 17092020
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lung Hernia; Thoracoscopy; Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During patient follow up the investigators noticed the occasional occurence of a lung herniation after uniportal Video assisted thoracoscopic surgery (VATS). Most of These patients were asymptomatic and didn't require any kind of treatment. To analyse the incidence of postoperative lung herniation after uniportal and the presence of symptoms the investigators decided to review every postoperative CT scan from January 2016 until March 2019 to radiologically identify postoperative lung herniations. Afterwards the investigators will contact the respective patient to ask for a follow-up physical examination and symptom evaluation (after consent was signed).

ELIGIBILITY:
Inclusion Criteria:

* Anatomical lung resection using uniportal VATS

Exclusion Criteria:

* Non anatomical lung resection
* Open surgery
* Pneumonectomy
* Informed consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient submitted to uniportal VATS anatomic lung resection from January 2016 until March 2019 who has had a postoperative radiological follow up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lung herniation | Postoperative follow-up up to 6 months
  Presence of intercostal lung herniation after uniportal VATS

SECONDARY OUTCOMES:
Symptoms | Postoperative follow-up to 5 years
  Symptoms described by patients presenting an intercostal lung hernia
Risk factors | At the time of operation
  Presence of Risk factors associated with the development of intercostal lung hernia after uniportal VATS surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lutz, MD, Principal Investigator — Department of General Thoracic Surgery Bern University Hospital